CLINICAL TRIAL: NCT04086706
Title: Retroflexion In The Ascending Colon Is A Costless Endoscopic Maneuver Increasing Adenoma Detection Rate
Status: Completed | Type: Observational
Sponsor: Alexandra Hospital, Athens, Greece (Other)
Responsible Party: Principal Investigator, SPYRIDON MICHOPOULOS, Head of GI Department, PhD, MD, Alexandra Hospital, Athens, Greece
Other Study IDs: AlexandraHospital
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Colonoscopy; Adenoma Detection Rate; Adenoma Miss Rate; Retroflexion
Keywords: Colonoscopy; Retroflexion; Adenoma Detection Rate; Adenoma Miss Rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Consecutive Patients with complete colonoscopy: Inclusion criteria were as follows: Patients older than 18 years, with a complete colonoscopy, for CRC screening or post-polypectomy surveillance or diagnostic assessment. Exclusion criteria precluded patients with previous colectomy or an abdominal surgery in the last 6 months, patients with polyposis syndromes or inflammatory bowel diseases and if they were unfit for polypectomy or the polyp specimen was not retrieved for histology.
  Interventions: Procedure: Retroflexion in the Right Colon

INTERVENTIONS:
Procedure: Retroflexion in the Right Colon — Prospective evaluation of an every day technique (retroflexion) used in our department for many years. The protocol of ascending colon examination encompassed 2 phases: A first phase (1) divided in Forward view (1a) videlicet insertion from the right flexure to the caecum followed by a second forward view (1b) namely withdrawal till the right flexure and reinsertion to the caecum maintaining the endoscope straight and a second phase (2, Retroflexion) with U-turn of the colonoscope in the caecum till the right flexure and then redressing to the forward view and reinsertion to the caecum.

SUMMARY:
Missing polyps during colonoscopy is considered an important factor for interval cancer appearance especially in the ascending colon (AC). Aim of the study: To evaluate the contribution of retroflexion to adenoma detection in the AC. Patients-Methods: Prospective observational study included consecutive patients with complete colonoscopy between June 2017 and June 2018. The AC was examined in two phases. The first phase included two forward views from the hepatic flexure to the cecum and the second phase a retroflexion in the cecum, inspection till the hepatic flexure then redressing to forward view and reinsertion to the cecum.

DETAILED DESCRIPTION:
We prospectively evaluated for polyp detection in the ascending colon a cohort of consecutive patients addressed (intended) for complete colonoscopy in Alexandra University Hospital, Athens, Greece for a predetermined period (June 2017-June 2018). All colonoscopies were performed under conscious sedation by using midazolam and/or propofol and continuous monitoring for vital signs. The type of endoscopes used were adult high definition, with variable stiffness, colonoscopes Olympus Evis Exera CF-H185 and 190. Insufflation was performed by means of a CO2 insufflator (OLYMPUS - UCR). An irrigation pump (OLYMPUS - OFP2) was used if needed, either for washing or for water exchange technique according to the endoscopist judgement. Oral sodium and potassium sulphate in combination (Eziclen®) or PEG solutions (Klean Prep® or Fortrans®) were used for bowel preparation which was measured by means of the Segmental Boston Bowel Preparation Scale. Inclusion criteria were as follows: Patients older than 18 years, with a complete colonoscopy, for CRC screening or post-polypectomy surveillance or diagnostic assessment. Exclusion criteria precluded patients with previous colectomy or an abdominal surgery in the last 6 months, patients with polyposis syndromes or inflammatory bowel diseases and if they were unfit for polypectomy or the polyp specimen was not retrieved for histology. The protocol of ascending colon examination encompassed 2 phases: A first phase (1) divided in Forward view (1a) videlicet insertion from the right flexure to the caecum followed by a second forward view (1b) namely withdrawal till the right flexure and reinsertion to the caecum maintaining the endoscope straight and a second phase (2, Retroflexion) with U-turn of the colonoscope in the caecum till the right flexure and then redressing to the forward view and reinsertion to the caecum.

Concerning endoscopy 2 seniors and 4 trainees participated in the study. All colonoscopies were performed with at least 2 operators, one senior and one trainee. The main investigator, the most experienced endoscopist in the department was present during all the procedures for the ascending colon examination (SM). Only 3 attempts were permitted for retroflexion achievement, performed by the main investigator if a younger trainee or senior gastroenterologist could not perform it. Polyps were mapped during both phases and were not removed until the end of the inspection. Polypectomy followed according to the previous mapping and all polyps were collected and sent for histological examination. The protocol of this non-interventional study as well as the informed consent for the patients were submitted and approved by the local ethical committee.

Adenoma detection rate (ADR) was defined as the number of colonoscopies in which one or more adenomas were detected, divided by the total number of colonoscopies. ADR in the ascending colon as the number of colonoscopies with at least one adenoma in the ascending colon divided by the total number of colonoscopies. Adenoma miss rate (AMR) of the ascending colon was defined as the number of additional adenomas in ascending colon detected by retroflexed view divided by the total adenomas in ascending colon detected with two forward and retroflexion views. The per-patient miss rate was calculated as the number of patients with additional adenomas detected on retroflexion divided by the total number of patients who underwent the examination.

Finally we evaluated two additional quality parameters in order to assess the contribution of retroflexion in adenoma detection: adenomas per colonoscopy (APC) calculated by dividing the number of detected adenomas by the total number of colonoscopies and adenomas per positive participant (APP) calculated by dividing the number of detected adenomas by the number of colonoscopies in which at least 1 adenoma was detected.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients with a complete colonoscopy
* Patients with indication for colonoscopy of CRC screening, post-polypectomy surveillance or diagnostic assessment

Exclusion Criteria:

* patients with previous colectomy or an abdominal surgery in the last 6 months
* patients with polyposis syndromes
* patients inflammatory bowel diseases
* patients unfit for polypectomy
* if the polyp specimen was not retrieved for histology

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: consecutive patients intended for complete colonoscopy in Alexandra University Hospital, Athens, Greece for a predetermined period (June 2017-June 2018) were prospectively evaluated for polyp detection in the ascending colon
Sampling Method: Non-Probability Sample
Enrollment: 655 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Adenoma Miss Rate | June 2017-June 2018
  adenoma miss rate by performing systematically a retroflexion after a second forward view in the ascending colon and evaluate the additional gain in adenoma detection
Increase in Adenoma Detection Rate in the ascending Colon | June 2017-June 2018
  adenoma miss rate by performing systematically a retroflexion after a second forward view in the ascending colon and evaluate the additional gain in adenoma detection

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandra General Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Desai M, Bilal M, Hamade N, Gorrepati VS, Thoguluva Chandrasekar V, Jegadeesan R, Gupta N, Bhandari P, Repici A, Hassan C, Sharma P. Increasing adenoma detection rates in the right side of the colon comparing retroflexion with a second forward view: a systematic review. Gastrointest Endosc. 2019 Mar;89(3):453-459.e3. doi: 10.1016/j.gie.2018.09.006. Epub 2018 Sep 14. PMID 30222971
- [Background] Triantafyllou K, Tziatzios G, Sioulas AD, Beintaris I, Gouloumi AR, Panayiotides IG, Dimitriadis GD. Diagnostic yield of scope retroflexion in the right colon: A prospective cohort study. Dig Liver Dis. 2016 Feb;48(2):176-81. doi: 10.1016/j.dld.2015.11.024. Epub 2015 Dec 2. PMID 26748425
- [Background] Kim HU, Boo SJ, Na SY, Song HJ. [Additional polyp detection rate using colonoscopic retroflexion in right colon]. Korean J Gastroenterol. 2015 Feb;65(2):90-8. doi: 10.4166/kjg.2015.65.2.90. Korean. PMID 25716711
- [Background] Hewett DG, Rex DK. Miss rate of right-sided colon examination during colonoscopy defined by retroflexion: an observational study. Gastrointest Endosc. 2011 Aug;74(2):246-52. doi: 10.1016/j.gie.2011.04.005. Epub 2011 Jun 15. PMID 21679946
- [Background] Harrison M, Singh N, Rex DK. Impact of proximal colon retroflexion on adenoma miss rates. Am J Gastroenterol. 2004 Mar;99(3):519-22. doi: 10.1111/j.1572-0241.2004.04070.x. PMID 15056095
- [Background] Chandran S, Parker F, Vaughan R, Mitchell B, Fanning S, Brown G, Yu J, Efthymiou M. Right-sided adenoma detection with retroflexion versus forward-view colonoscopy. Gastrointest Endosc. 2015 Mar;81(3):608-13. doi: 10.1016/j.gie.2014.08.039. Epub 2014 Oct 29. PMID 25440687
- [Background] Lee HS, Jeon SW, Park HY, Yeo SJ. Improved detection of right colon adenomas with additional retroflexion following two forward-view examinations: a prospective study. Endoscopy. 2017 Apr;49(4):334-341. doi: 10.1055/s-0042-119401. Epub 2016 Dec 8. PMID 27931050